CLINICAL TRIAL: NCT02516696
Title: Lenalidomide and Dexamethasone (Rd) Versus Clarithromycin [Biaxin®] / Lenalidomide [Revlimid®] / Dexamethasone (BiRd) as Initial Therapy in Multiple Myeloma
Brief Title: BiRd vs. Rd as Initial Therapy in Multiple Myeloma
Acronym: BiRd vs Rd
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1411015662; RV-CL-MM-PI-004078 (Other Grant/Funding Number: Celgene Corporation)
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Clarithromycin; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BiRD treatment regimen (Experimental): Subjects on the BiRD arm will receive clarithromycin, lenalidomide, and dexamethasone in 28-day cycles.
  Interventions: Drug: Clarithromycin; Drug: Lenalidomide; Drug: Dexamethasone
- Rd treatment regimen (Active Comparator): Subjects on the Rd arm will receive lenalidomide and dexamethasone in 28-day cycles.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Clarithromycin — 500mg PO twice daily on days 1-28 for a 28-day cycle.
  Other Names: biaxin
  Arms: BiRD treatment regimen
Drug: Lenalidomide — 25 mg PO days 1-21 followed by a 7 day rest period for each 28-day cycle
  Other Names: Revlimid
Drug: Dexamethasone — 20 mg PO on Days 1, 8, 15, and 22 for each cycle for subjects 75 years and younger.
  Other Names: Decadron

SUMMARY:
This is a randomized, open-label, phase III study to investigate the efficacy of combination therapy with an induction phase utilizing a combination clarithromycin (Biaxin®), lenalidomide (Revlimid®), dexamethasone (Decadron®), in multiple myeloma patients who are newly diagnosed and require treatment when compared to patients who receive lenalidomide and dexamethasone alone.

DETAILED DESCRIPTION:
This research study is for men and women with newly diagnosed, previously untreated multiple myeloma. The purpose of this study is to observe the how well the different combinations of study drugs work as therapy for patients with newly diagnosed, transplant ineligible, previously untreated multiple myeloma.

The study will be done in two arms:

BiRd Arm:

* Clarithromycin 500mg PO twice daily on days 1-28 for a 28-day cycle
* Lenalidomide 25mg PO daily on days 1-21 of a 28-day cycle
* Dexamethasone 40mg PO will be given on days 1, 8, 15, 22 of a 28-day cycle

Rd Arm:

* Lenalidomide 25mg PO daily on days 1-21 of a 28-day cycle
* Dexamethasone 40mg PO will be given on days 1, 8, 15, 22 of a 28-day cycle

Subjects will be treated in 28-day cycles and may continue treatment as long as they are responding to therapy and not experiencing unacceptable side effects or disease progression. There will be an evaluation at the end of each cycle. Participants will be in the study until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily sign and understand written informed consent.
* Subject is at least 65 years old at the time of signing the consent form.
* Subject has histologically confirmed multiple myeloma that has never before been treated
* Subject has no prior anti-myeloma treatment therapy within 14 days prior to initiation of study treatment except for corticosteroids with a maximum allowed dosage equivalent to three pulses of dexamethasone (40mg daily for 4 days equals one pulse). Patients may have received prior adjuvant antiresorptive therapy (i.e., pamidronate or zoledronic acid) as routine care, or radiation therapy as palliation for pain and/or spinal cord compression.
* Subject has measurable disease as defined by > 0.5 g/dL serum monoclonal protein, >10 mg/dL involved serum free light chain (either kappa or lambda) provided that the serum free light chain ratio is abnormal, >0.2 g/24 hrs urinary M-protein excretion, and/or measurable plasmacytoma(s) of at least 1cm in greatest dimension as measured by either CT scanning or MRI.
* Subject has a Karnofsky performance status ≥60% (>50% if due to bony involvement of myeloma (see Appendix IV).
* Subject is able to take prophylactic anticoagulation as detailed in section 9.1 (patients intolerant to aspirin may use warfarin or low molecular weight heparin).
* Subject is registered into the mandatory RevAssist® program, and is willing and able to comply with the requirements of RevAssist® program.
* If subject is a female of childbearing potential (FCBP),† she must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide
* Subject has a life expectancy ≥ 3 months
* Subjects must meet the following laboratory parameters:

  * Absolute neutrophil count (ANC) ≥750 cells/mm3 (1.0 x 109/L)
  * Hemoglobin ≥ 7 g/dL
  * Platelet count ≥ 30,000/mm3 (75 x 109/L)
  * Serum SGOT/AST <3.0 x upper limits of normal (ULN)
  * Serum SGPT/ALT <3.0 x upper limits of normal (ULN)
  * Serum total bilirubin <2.0 mg/dL (34 µmol/L)
  * Creatinine clearance ≥ 45 cc/min

Exclusion Criteria:

* Subject has immeasurable MM (no measurable monoclonal protein, free light chains in blood or urine, or measureable plasmacytoma on radiologic scanning).
* Subject has a prior history of other malignancies unless disease free for ≥ 5 years, except for basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or localized prostate cancer with Gleason score < 7 with stable prostate specific antigen (PSA) levels.
* Subject has had myocardial infarction within 6 months prior to enrollment , or NYHA(New York Hospital Association) Class III or IV heart failure (see APPENDIX VI), Ejection Fraction < 35%, uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Female subject who is pregnant or lactating.
* Subject has known HIV infection
* Subject has known active hepatitis B or hepatitis C infection.
* Subject has active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program.
* Subject is unable to reliably take oral medications
* Subject has known hypersensitivity to dexamethasone, clarithromycin, lenalidomide, or thalidomide
* Subject has a history of thromboembolic event within the past 4 weeks prior to enrollment.
* Subject has any clinically significant medical or psychiatric disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.
* Subject has previously been treated for multiple myeloma

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Monge, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - University of Colorado - Anschutz Cancer Center, Aurora, Colorado
  - Weill Cornell Medical College, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BiRD Treatment Regimen | Rd Treatment Regimen
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BiRD Treatment Regimen | Rd Treatment Regimen | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 7 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 4 | 11
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Survival Duration Without Disease Progression
Description: Calculate rate of progression-free survival for subjects following treatment BiRd regimen compared to Rd treatment regimen. Progression is determined by the International Myeloma Working Group Criteria.
Time Frame: Until disease progression or death from any cause, for a maximum of approximately 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BiRD Treatment Regimen | Rd Treatment Regimen
Number analyzed (Participants) | 7 | 5
days | 661 [586 to NA] — Some participants were still alive without disease progression at the time of study completion. | 1694 [821 to NA] — Some participants were still alive without disease progression at the time of study completion.

2. Secondary Outcome: Overall Response Rate
Description: Capture the number of subjects who demonstrate a complete or partial response to treatment with BiRD regimen, as compared to Rd. Complete and partial responses are defined by the International Myeloma Working Group Criteria.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | BiRD Treatment Regimen | Rd Treatment Regimen
Number analyzed (Participants) | 7 | 5
Participants | 7 | 4

3. Secondary Outcome: Number of Adverse Events Experienced
Description: Capture the number of adverse events experienced with BiRd regimen as compared to Rd regimen
Time Frame: 2 years
Measure: Number; unit: adverse events
Arm/Group | BiRD Treatment Regimen | Rd Treatment Regimen
Number analyzed (Participants) | 7 | 5
adverse events | 79 | 67

4. Secondary Outcome: Overall Survival
Description: Survival following treatment to the date of death of subjects on BiRd regimen as compared to Rd.
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BiRD Treatment Regimen | Rd Treatment Regimen
Number analyzed (Participants) | 7 | 5
days | NA [906 to NA] — Median overall survival was not reached for patients in the BiRd arm (95% CI: 906-NA). | 1014 [821 to NA] — Participants were still alive at the time of study closure.

5. Secondary Outcome: Number of Days After Initiating Treatment With BiRd Regimen to Disease Progression, as Compared to Subjects on Rd Treatment Regimen.
Description: Progression is determined by the International Myeloma Working Group Criteria.
Time Frame: Until disease progression for a maximum of approximately 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BiRD Treatment Regimen | Rd Treatment Regimen
Number analyzed (Participants) | 7 | 5
days | 661 [661 to NA] — Not all participants progressed at the time of study completion. | 1694 [NA to NA] — Not all participants progressed at the time of study completion.

6. Secondary Outcome: Number of Patients With Objective Response Rate (CR+PR)
Time Frame: up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | BiRD Treatment Regimen | Rd Treatment Regimen
Number analyzed (Participants) | 7 | 5
Participants | 7 | 4

7. Secondary Outcome: Number of Patients With Complete Response Rate (CR)
Description: Complete response is defined by the International Myeloma Working Group Criteria.
Time Frame: up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | BiRD Treatment Regimen | Rd Treatment Regimen
Number analyzed (Participants) | 7 | 5
Participants | 2 | 0

8. Secondary Outcome: Number of Days for Event-Free Survival
Description: Descriptively presented for each treatment group and no formal statistical comparison will be made between treatment arms
Time Frame: approximately 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BiRD Treatment Regimen | Rd Treatment Regimen
Number analyzed (Participants) | 7 | 5
days | 336 [225 to NA] — Not all patients progressed by the time of study completion. | 821 [310 to NA] — Not all patients progressed by the time of study completion.

9. Secondary Outcome: Number of Days for Duration of Response
Description: as for outcome 8
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BiRD Treatment Regimen | Rd Treatment Regimen
Number analyzed (Participants) | 7 | 5
days | 308 [227 to NA] — Some participants continued to have a sustained response at the time of study completion. | 803 [282 to NA] — Some participants continued to have a sustained response at the time of study completion.

10. Secondary Outcome: Number of Months to Progression-Free Survival 2
Description: Time from study entry until 2nd instance of disease progression. Progression is determined by the International Myeloma Working Group Criteria. Descriptively presented for each treatment group and no formal statistical comparison will be made between treatment arms.
Time Frame: approximately 5 years
Population: Data not collected due to early trial termination due to low accrual.
Arm/Group | BiRD Treatment Regimen | Rd Treatment Regimen
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue Subscale (FS; Version 4) Score of Patients Receiving BiRd vs Rd Treatment
Description: The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a 40-item measure that assesses self-reported fatigue and its impact upon daily activities and function. The FACIT- Fatigue Subscore (FS) is comprised of 13 items, within the total 40-item FACIT-F, that assess fatigue and its impact. This analysis is only based on the FS score. Items are scored on a 5 point Likert-type scale. Item scores can range from 0 ("not at all") to 4 ("very much"), and the total, summed score from 0 to 52; lower scores indicate greater fatigue. The recall period for each item is the past 7 days. Data is descriptively presented for each treatment group and no formal statistical comparison will be made between treatment arms.
Time Frame: up to 3 years
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | BiRD Treatment Regimen | Rd Treatment Regimen
Number analyzed (Participants) | 7 | 2
Score on a scale | 32.75 [16.9 to 45.46] | 37.24 [28.58 to 45.89]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent until participants were removed from the study, or for a maximum of 60 months. Participants were removed at the time of disease progression, death, or study termination, whichever occurred first. This study was terminated early due to low accrual.
Arm/Group | BiRD Treatment Regimen | Rd Treatment Regimen
All-Cause Mortality (participants affected / at risk) | 2/7 | 4/5
Serious Adverse Events (participants affected / at risk) | 6/7 | 3/5
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BiRD Treatment Regimen (N=7) | Rd Treatment Regimen (N=5)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Allergic Reaction (General disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Fall (General disorders) | 2 (3) | 1 (1)
Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Syncope (General disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Secondary Primary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (3)
Edema Limbs (General disorders) | 0 (0) | 1 (1)
Skin Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
COVID-19 Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BiRD Treatment Regimen (N=7) | Rd Treatment Regimen (N=5)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hyponatremia (Investigations) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Decreased albumin (Investigations) | 1 (1) | 0 (0)
Increased alkaline phosphatase (Investigations) | 1 (1) | 0 (0)
Anorexia (General disorders) | 1 (1) | 2 (3)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Cold Symptoms (General disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 2 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (3)
Fall (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (6) | 2 (2)
Hair loss (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Hypertension (Investigations) | 1 (1) | 0 (0)
Hypocalcemia (Investigations) | 2 (3) | 1 (1)
Hypokalemia (Investigations) | 0 (0) | 1 (1)
Hypomagnesemia (Investigations) | 1 (1) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 1 (1)
Dysgeusia (General disorders) | 1 (1) | 1 (1)
Leukocytosis (Investigations) | 1 (1) | 0 (0)
Leukopenia (Investigations) | 1 (1) | 1 (1)
Edema Limbs (General disorders) | 2 (3) | 2 (2)
Pain (General disorders) | 2 (4) | 2 (4)
Lymphopenia (Investigations) | 1 (3) | 0 (0)
Maculo-papular rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral Neuropathy (Nervous system disorders) | 1 (1) | 1 (2)
Post-nasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin Atrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Investigations) | 2 (3) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal Yeast Infection (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Weight Loss (General disorders) | 0 (0) | 2 (2)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Allergic Rhinitis (General disorders) | 0 (0) | 1 (1)
Body Aches (General disorders) | 0 (0) | 2 (2)
Bruising (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Dehydration (General disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Gun sensitivity/inflammation (General disorders) | 0 (0) | 1 (1)
Extremity Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lower extremity weakness (General disorders) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 1 (1)
Mucosal Infection/Thrush (Infections and infestations) | 0 (0) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The significance of these results is limited by the study's low accrual. The study's low accrual was due in part to the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT02516696/Prot_SAP_000.pdf